CLINICAL TRIAL: NCT05669846
Title: Phase II Feasibility Study of Healthy Donor FMT (hdFMT) and Pembrolizumab in Relapsed/Refractory (R/R) PD-L1 Positive NSCLC
Brief Title: Study of Healthy Donor FMT (hdFMT) and Pembrolizumab in Relapsed/Refractory (R/R) PD-L1 Positive NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Diwakar Davar (Other)
Collaborators: Gateway for Cancer Research (Other)
Responsible Party: Sponsor-Investigator, Diwakar Davar, Assistant Professor of Medicine - Hematology, Oncology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 22-078
Record Dates: First submitted 2022-12-20; First posted 2023-01-03 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Relapsed; Refractory; Healthy Donor FMT (hdFMT)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Recurrence | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Healthy Donor Fecal Microbiota Transplant (hdFMT) with Pembrolizumab (Experimental): The hdFMT along with an intestinal biopsy will be performed as outpatient by a gastroenterologist. The hdFMT is infused into the colon by performing a colonoscopy (Treatment Phase 1) and by a sigmoidoscopy or oral capsules (Treatment Phase 2). FMT will be performed on Cycle 1 Day 1 and Cycle 3 Day 1 during Treatment Phase 1 and every 9 weeks starting with Cycle 4 Day 1 during Treatment Phase 2.
  Pembrolizumab, 200mg, will be administered as a 30-minute IV infusion every 3 weeks starting Cycle 1 Day 1 (same day as the hdFMT), and continue on Day 1 of each 21-day cycle.
  Interventions: Drug: Healthy Donor Fecal Microbiota Transplant (hdFMT); Drug: Pembrolizumab

INTERVENTIONS:
Drug: Healthy Donor Fecal Microbiota Transplant (hdFMT) — FMT is a procedure in which fecal matter or stool is collected from a tested donor, mixed with a saline or other solution, strained and infused into the colon by performing a colonoscopy and sigmoidoscopy, or, administered orally in the form of capsules. The FMT consists of introducing normal bacterial flora contained in the stool collected from a healthy donor into the small intestine. In this case, the hdFMT will be administered on Cycle 1 Day 1 and Cycle 3 Day 1 during Treatment Phase 1 and every 9 weeks starting with Cycle 4 Day 1 during Treatment Phase 2.
Drug: Pembrolizumab — Pembrolizumab, 200mg, will be administered as a 30-minute IV infusion every 3 weeks starting Cycle 1 Day 1 (same day as the FMT), and continue on Day 1 of each 21-day cycle.
  Other Names: Keytruda

SUMMARY:
This study is to determine if Healthy Donor FMT (hdFMT) improves the body's ability to fight cancer in patients with relapsed/refractory PD-L1 Positive NSCLC.

DETAILED DESCRIPTION:
The study evaluating the addition of Healthy Donor FMT (hdFMT) to pembrolizumab in PD-1 R/R NSCLC will be conducted over a 104-week period. Patients with anti-PD-1 R/R NSCLC are eligible to enroll. Prior exposure to microbiome modulating therapy is exclusionary. Suitable patients will be identified at the time of progression upon PD-1 monotherapy or PD-1 containing regimens. Patients will undergo a 35-day screening evaluation consisting of systemic staging scans, tumor biopsy, stool/blood serologic studies to confirm suitability.

Once enrolled, patients will be seromatched with a suitable donor. Suitable donors are advanced cancer patients who have undergone PD-1 monotherapy and are currently in durable remission (median PFS >24 months from initiation of PD-1 therapy) with no ongoing irAE as delineated below. Patients will receive Healthy Donor FMT (hdFMT) (induction) via colonoscopy on C1D1 and C3D1. R-FMT (maintenance) via sigmoidoscopy on C4D1 and will be repeated every 9 weeks. All patients will additionally receive pembrolizumab at 200mg every three weeks. Patients will be treated until disease progression or intolerable toxicity or completion of 2 years of therapy, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

Male participants:

• A male participant must agree to use a contraception as detailed per protocol of this protocol during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.

* Female participants:

  • A female participant is eligible to participate if she is not pregnant per protocol, not breastfeeding, and at least one of the following conditions applies:
  * Not a woman of childbearing potential (WOCBP); OR
  * A WOCBP who agrees to follow the contraceptive guidance per protocol during the treatment period and for at least 120 days after the last dose of study treatment.
* Histologically or cytologically confirmed diagnosis of stage IV PD-L1+ NSCLC.

  * NOTE: Patients with either squamous or non-squamous NSCLC may enroll.
  * NOTE: Documented PD-L1 status (defined as 1% or greater) as determined by immunohistochemistry with anti-PD-L1 antibody (IHC 22C3 pharmDx or other FDA approved diagnostic method) from a core or excisional biopsy (fine needle aspirate is not sufficient).
  * NOTE: Patients with small cell, large cell, neuroendocrine and/or sarcomatoid NSCLC are excluded.
* Participants must have progressed on treatment with an anti-PD(L)1 ICI administered either as monotherapy or in combination with other checkpoint inhibitors or other standard/investigational therapies. PD-1 treatment progression is defined by meeting all the following criteria:

  * Has received at least 2 doses of an approved anti-PD(L)1 ICI administered as a single agent, in combination with chemotherapy, and/or in combination with other investigational therapy.
  * Participants who progressed on/within 3 months of adjuvant therapy with anti-PD(L)1 ICI will eligible.
  * Demonstrated disease progression after anti-PD-1/L1 as defined by RECIST v1.1. The initial evidence of PD is to be confirmed by a second assessment no sooner than 4 weeks from the date of the first documented PD.
  * Progressive disease has been documented within 12 weeks from the last dose of anti-PD-1/anti-PD-L1 mAb.
  * NOTE: Progressive disease must be determined as above.
  * NOTE: This determination is made by the treating investigator. Once PD is confirmed, the initial date of PD documentation will be considered the date of PD.
  * NOTE: Anti-PD(L)1 ICI need not be the most recent line of therapy administered.
* Patients with CNS disease are eligible if CNS metastases are treated and deemed stable prior to date of enrollment.

  * NOTE: All patients will undergo CNS imaging at the time of Screening. Patients with treated brain metastases will need repeat CNS imaging to document stability.
  * NOTE: Stability is defined based on appearance of treated lesions on a contrast-enhanced CT or MRI brain study performed as part of screening by radiologist, radiation oncologist or neurosurgeon (whichever is most appropriate); absence of new or enlarging brain metastases; and no longer requiring systemic steroids (≤ 10 mg/day prednisone or equivalent) for at least one week prior to enrollment.
  * NOTE: The contrast-enhanced CT or MRI brain imaging study should be performed no sooner than 2 weeks after most recent surgical and/or radiological intervention.
  * NOTE: If lesions were discovered during Screening, the patient may be eligible if the lesions are treated and stable based on the above criteria.
  * NOTE: Patients with leptomeningeal involvement (leptomeningeal enhancement on MRI/CT imaging and/or positive CSF cytology) are excluded regardless of stability.
* Prior treatment(s)

  * NOTE: Prior anti-CTLA-4 ICI is allowed but not required.
  * NOTE: Patients with known oncogenic driver (including but not limited to EGFR, ALK, ROS, MET alterations) must have received and progressed past driver-specific therapy
* Willingness to repeatedly receive FMT administered endoscopically (colonoscopy or sigmoidoscopy) and via pills following necessary bowel preparation pre-procedure.

  * NOTE: Understands infectious risks associated with FMT administration. o Although FMT infusate has been screened for bacteria, viruses, fungi and parasites there is a risk of transmission of known and unknown infectious organisms contained in the donor stool. Post-FMT bacteremia (e.g. E. coli), sepsis and fatal events may rarely occur.
  * NOTE: Understands non-infectious risks associated with FMT administration. o Possible allergy and/or anaphylaxis to antigens in donor stool.

    o Theoretical risk of developing disease possibly related to donor gut microbiota including but not limited to: obesity, metabolic syndrome, cardiovascular disease, autoimmune conditions, allergic/atopic disorders, neurologic disorders, psychiatric conditions and malignancy.
  * NOTE: Understand risks associated with endoscopy (colonoscopy or sigmoidoscopy) including risk of infection transmission, colonic perforation, aspiration pneumonia, and death.
  * NOTE: Understand that data regarding the long-term safety risk of FMT are lacking.
* Presence of measurable disease based on RECIST 1.1.

  * Patients need to have at least one measurable lesion and a separate lesion for biopsy. Patients with only 1 lesion may be enrolled after discussion with Sponsor-Investigator.
  * Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Able to provide newly obtained core or excisional biopsy of a tumor lesion not previously irradiated to undergo tumor biopsy (core, punch, incisional or excisional).

  • Biopsy must meet minimal sampling criteria as defined per protocol.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Have adequate organ function per protocol. Specimens must be collected within 28 days prior to the start of study intervention.
* Criteria for patients with hepatitis B and C

  * Screening for hepatitis B and C are required.
  * For hepatitis B positive patients:

    * Patients who are hepatitis B positive (i.e. HBsAg positive) or have a history of history of hepatitis B (i.e. HBcAb positive, or history of documented hepatitis B infection) are eligible if they have received hepatitis B directed antiviral therapy for at least 4 weeks and have undetectable HBV viral load (HBV DNA) prior to enrollment.
    * Participants should remain on antiviral therapy throughout study intervention and follow local guidelines for HBV antiviral therapy post completion of study intervention.
  * For hepatitis C positive patients:

    * Patients who are hepatitis C positive (i.e. HCV antibody reactive) or have a history of history of hepatitis C (i.e. history of documented hepatitis C infection) are eligible if they have received and completed hepatitis C directed antiviral therapy at least 4 weeks and have undetectable HCV viral load (HCV RNA) prior to enrollment.

Exclusion Criteria:

* Diagnosis of NSCLC histologies other than squamous and/or adenocarcinoma histologies including small cell, large cell, neuroendocrine and/or sarcomatoid histologies.
* Prior therapies:

  * Receipt of prior agent(s) targeting the intestinal microbiome including but not limited to: FMT, defined bacterial consortia, single bacterial species and/or microbiota derived peptides.
  * Prior chemotherapy, targeted therapy, and/or small molecule therapy within 2 weeks (or 4 half lives) prior to study Day 1.
  * Prior radiotherapy within 2 weeks of start of study intervention.

    * Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.
    * A 2-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to disease including CNS disease.
* Presence of an absolute contraindication(s) to FMT administration

  • Toxic megacoon
  * Severe dietary allergies (e.g. shellfish, nuts, seafood)
  * Inflammatory bowel disease
* Patients who have not adequately recovered (i.e., ≤Grade 1 or at baseline or ≤Grade 2 endocrinopathy) from adverse events (AEs) due to a previously administered agent.
* A WOCBP who has a positive urine pregnancy test at Screening (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Has received a live vaccine within 30 days prior to the first dose of study drug.

  * Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), SARS-CoV-2 and typhoid vaccine.
  * Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 14 days prior to the first dose of study drug.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).

  • NOTE: Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
* Concurrent non-hematologic malignancy within 3 years of data of first planned dose of therapy except for tumors with a negligible risk of metastasis and/or death as defined below:

  * Adequately treated non-invasive malignancies including but not limited to melanoma in situ (MIS), cutaneous squamous cell carcinoma (cSCC), in situ cSCC, basal cell carcinoma (BCC), CIS of cervix, or DCIS/LCIS of breast.
  * Low-risk early-stage prostate adenocarcinoma (T1-T2a N0 M0 and Gleason score ≤6 and PSA ≤10 ng/mL) for which the management plan is active surveillance, or prostate adenocarcinoma with biochemical-only recurrence with documented PSA doubling time of > 12 months for which the management plan is active surveillance.
  * Indolent hematologic malignancies for which the management plan is active surveillance including but not limited to CLL/indolent lymphoma.

    * Patients with high-risk hematologic malignancies (CML, ALL, AML, Hodgkin's or non-Hodgkin's lymphoma) are excluded even if the management plan is active surveillance.
* Active (i.e., symptomatic or growing) central nervous system (CNS) metastases.

  * NOTE: Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 2 weeks by repeat imaging (note that the repeat imaging should be performed during Screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention as delineated in Section 4.1.7.
  * NOTE: Patients with leptomeningeal disease are excluded.
* Has severe hypersensitivity (≥Grade 3) to anti-PD(L)1 inhibitor.
* Has a systemic disease that requires systemic pharmacologic doses of corticosteroids greater than 10 mg daily prednisone (or equivalent).

  * NOTE: Participants who are currently receiving steroids at a dose of ≤10 mg daily do not need to discontinue steroids prior to enrollment.
  * NOTE: Participants that require topical, ophthalmologic, injected and/or inhalational steroids are not excluded from the study.
  * NOTE: Participants with hypothyroidism stable on hormone replacement or Sjogren's syndrome are not excluded from the study.
  * NOTE: Participants who require active immunosuppression (greater than steroid dose discussed above) for any reason are excluded from the study.
* Has a history of interstitial lung disease or active, non-infectious pneumonitis that required steroids or has current pneumonitis.
* Has a history of non-infectious myocarditis or symptomatic cardiac co-morbidities requiring active management.

  * NOTE: Patients with a history of symptomatic congestive heart failure (New York Heart Association Functional Classification III or IV) are excluded.
  * NOTE: Patients with a history of unstable angina, serious uncontrolled cardiac arrhythmia, or myocardial infarction 6 months prior to study entry are excluded.
* Active infections

  * Any active infection requiring systemic therapy.
  * Active TB (Bacillus Tuberculosis).
  * Active COVID-19 infection and/or exposure to SARS-CoV-2 as defined below:

    * Positive SARS-CoV-2 result on nasopharyngeal (by RT-PCR test)
    * Active COVID-19 infection (per CDC guidelines)
    * Exposure to active COVID-19 infected patient (as confirmed using SARS-CoV-2 RT-PCR test or other approved test) as defined per CDC guidelines.
  * Active human immunodeficiency virus (HIV) infection.

    o Patients will be evaluated for HIV during screening.
  * Concurrent active Hepatitis B (defined as HBsAg positive and/or detectable HBV DNA) and Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the Screening visit through 120 days after the last dose of trial treatment.
* Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) per RECIST v1.1 | Up to 5 years
  The proportion of patients with objective response (Complete Response (CR) or Partial Response (PR)) to R-FMT and pembrolizumab treatment in PD-1 primary refractory NSCLC as assessed per RECIST v1.1. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. For non-target lesions: Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10mm short axis); PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.

SECONDARY OUTCOMES:
Incidence of Adverse Events Related to Treatment | Up to 5 years
  Frequency of Adverse Events and specifically ≥grade 2 irAEs per CTCAE v5.0 in PD-1 primary refractory NSCLC in patients treated with Healthy Donor FMT (hdFMT) and pembrolizumab, to assess overall safety, feasibility and tolerability of treatment.
Objective Response Rate (ORR) per iRECIST | Up to 5 years
  The proportion of patients Complete Response (irCR) or Partial Response (irPR) to treatment as assessed per iRECIST. irCR:Disappearance of non-nodal lesions.All pathologic lymph nodes <10 mm (short axis) (2 consecutive measurements ≥4 weeks apart); irPR :≥30% decrease from baseline (2 consecutive measurements ≥4 weeks apart). Disappearance of all non-nodal lesions.All pathologic lymph nodes <10 mm (Non-Target Lesions:Any other than disappearance of all non-nodal lesions and reduction of pathologic lymph nodes <10 mm). Baseline tumor burden: sum of single diameters (short axis for nodal lesions, longest diameter for other lesions) for target lesions. In subsequent scans, the diameters of new measurable lesions are added to the tumor burden. Re-treatment: ≤5 target lesions (=/≠ original lesions) are selected and a new baseline tumor burden will be established. (no distinct iRECIST assessment until radiographic progression per RECIST 1.1 is observed).
CD8+ TIL and intra-tumoral myeloid cell density | Up to 5 years
  Percentage of CD8+ T cells in intra-tumoral myeloid cells in pre-treatment biopsy samples assess using multiplex IHC.
Progression-free Survival (PFS) | Up to 5 years
  The median length of time from initiation of study drug(s) disease progression as defined by RECIST v1.1, or death. Progressive Disease (PD): ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Overall Survival (OS) | Up to 5 years
  The median length of time that patients remain alive after treatment.
6-month Progression-free Survival | Up to 6 months
  Percentage of patients without disease progression at 6 months after start of treatment, per RECIST v1.1. Progressive Disease (PD): ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
1-year Progression-free Survival (PFS) | Up to 1 year
  Percentage of patients without disease progression at 1 year after start of treatment, per RECIST v1.1. Progressive Disease (PD): ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
2-year Progression-free Survival (PFS) | Up to 2 years
  Percentage of patients without disease progression at 2 years after start of treatment, per RECIST v1.1. Progressive Disease (PD): ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
1-year Overall Survival (OS) | Up to 1 year
  Percentage of patients that are alive at 1 year after start of treatment.
2-year Overall Survival (OS) | Up to 2 years
  Percentage of patients that are alive at 2 years after start of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Diwakar Davar, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No